CLINICAL TRIAL: NCT03400696
Title: Web-based Weight Loss Intervention
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: 23andMe, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: 23andMe_WLI001
Record Dates: First submitted 2018-01-04; First posted 2018-01-17 (Actual); Last update posted 2020-06-04 (Actual); Status verified 2020-06

CONDITIONS: Overweight and Obesity
Keywords: nutrition, diet, genetics, physical activity, weight loss
MeSH Terms: conditions — Overweight; Obesity; Motor Activity; Weight Loss

STUDY DESIGN:
Intervention Model Description: Participants are randomized to either a RCT or 'Participant choice' block, with 3 parallel interventions within each block
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- Randomized- Lower carbohydrate diet (Experimental)
  Interventions: Behavioral: Lower carbohydrate diet
- Randomized- Higher fiber diet (Experimental)
  Interventions: Behavioral: Higher fiber diet
- Randomized- Exercise focused (Experimental)
  Interventions: Behavioral: Physical activity focused
- Participant chooses- Lower carbohydrate diet (Experimental)
  Interventions: Behavioral: Lower carbohydrate diet
- Participant chooses- Higher fiber diet (Experimental)
  Interventions: Behavioral: Higher fiber diet
- Participant chooses- Exercise focused (Experimental)
  Interventions: Behavioral: Physical activity focused

INTERVENTIONS:
Behavioral: Lower carbohydrate diet — Focused on limiting dietary carbohydrates, eating healthy fat and protein sources, and engaging in physical activity
  Arms: Participant chooses- Lower carbohydrate diet; Randomized- Lower carbohydrate diet
Behavioral: Higher fiber diet — Focused on increasing dietary fiber, lowering fat intake from animal sources, and engaging in physical activity
  Arms: Participant chooses- Higher fiber diet; Randomized- Higher fiber diet
Behavioral: Physical activity focused — Focused on aerobic and resistance exercise, while following dietary guidelines <https://www.choosemyplate.gov>
  Arms: Participant chooses- Exercise focused; Randomized- Exercise focused

SUMMARY:
Excess weight is a major risk factor underlying leading causes of death globally, including cardiovascular disease, type 2 diabetes, and some cancers. Among participants assigned to the same lifestyle intervention arms in prior weight loss randomized controlled trials, large inter-individual differences in weight loss success have been observed, ranging from >50lbs of weight loss to >10lbs of weight gain. Both genetic and non-genetic factors underlying differential adherence and weight loss success are poorly understood.

DETAILED DESCRIPTION:
23andMe aims to recruit 91,227 adults to participate in a web-based weight loss intervention. Primary aims include: a.) to confirm whether AG/GG individuals at MTIF3 rs1885988 lose more weight on lifestyle interventions; and b.) to test the performance of a randomized controlled trial vs. self-selection study design in terms of weight loss, drop-outs, and adherence. Secondary (exploratory) analyses will focus on discovery of genetic and non-genetic predictors of weight loss success overall, and examination of potential interactions by intervention type. Web-administered intervention content, videos, and forums will be surfaced to participants every two weeks, and self-reported surveys will be surfaced weekly for the active intervention duration.

ELIGIBILITY:
Inclusion Criteria:

* US-based men and women in self-reported 'good' or better health
* Consented to participate in research
* BMI 25-40 kg/m2
* Not actively on a weight loss plan
* Willing and able to modify eating and physical activity patterns
* Not under a doctor's care for a serious medical condition

Exclusion Criteria:

* Are pregnant, lactating, within 6 months postpartum, or planning to become pregnant in the next 6 months
* Have diabetes (type 1 or 2) or are on hypoglycemic medications
* Had a heart attack or stroke within the past year
* Are unable or unwilling to follow a physical activity or diet intervention due to a medical condition or doctor's orders
* Have an eating disorder
* Have severe depression, anxiety, or other psychiatric conditions

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 63656 (Actual)
Dates: Start 2017-12-27 (Actual); Primary Completion 2019-01-08 (Actual); Study Completion 2019-04-16 (Actual)

PRIMARY OUTCOMES:
Change in weight from week 1 to week 12 of intervention | 12 weeks

SECONDARY OUTCOMES:
Change in waist circumference from week 1 to week 12 of intervention | 12 weeks
Change in waist-to-hip ratio from week 1 to week 12 of intervention | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Geoffrey Benton, PhD, Principal Investigator — 23andMe, Inc.; Liana Del Gobbo, PhD, Study Director — 23andMe, Inc.
Locations (1):
- 23andMe, Mountain View, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Papandonatos GD, Pan Q, Pajewski NM, Delahanty LM, Peter I, Erar B, Ahmad S, Harden M, Chen L, Fontanillas P; GIANT Consortium; Wagenknecht LE, Kahn SE, Wing RR, Jablonski KA, Huggins GS, Knowler WC, Florez JC, McCaffery JM, Franks PW; Diabetes Prevention Program and the Look AHEAD Research Groups. Genetic Predisposition to Weight Loss and Regain With Lifestyle Intervention: Analyses From the Diabetes Prevention Program and the Look AHEAD Randomized Controlled Trials. Diabetes. 2015 Dec;64(12):4312-21. doi: 10.2337/db15-0441. Epub 2015 Aug 7. PMID 26253612
- [Background] Bray MS, Loos RJ, McCaffery JM, Ling C, Franks PW, Weinstock GM, Snyder MP, Vassy JL, Agurs-Collins T; Conference Working Group. NIH working group report-using genomic information to guide weight management: From universal to precision treatment. Obesity (Silver Spring). 2016 Jan;24(1):14-22. doi: 10.1002/oby.21381. PMID 26692578